CLINICAL TRIAL: NCT02167243
Title: A Reinforcement Approach to Improve Diabetes Management - Randomized Trial
Brief Title: A Reinforcement Approach to Improve Diabetes Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1403013607; 1DP3DK097705-01 (NIH)
Record Dates: First submitted 2014-06-16; First posted 2014-06-19 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reinforcement for performing BG testing (Experimental): Subjects will receive reinforcement for BG testing. The intervention will reinforce subjects for conducting Self Monitoring of Blood Glucose (SMBG), with escalating reinforcers provided when subjects achieved sustained periods of testing at least 4 times/day at appropriate intervals.
  Interventions: Behavioral: Reinforcement for BG testing; Other: Standard of care
- No reinforcement for BG testing (Active Comparator): Subjects will receive standard of care without reinforcement for Self Monitoring Blood Glucose
  Interventions: Other: Standard of care

INTERVENTIONS:
Behavioral: Reinforcement for BG testing — Subjects will receive reinforcement for BG tests. The intervention will reinforce subjects for conducting Self Monitoring of Blood Glucose (SMBG), with escalating reinforcers provided when subjects achieved sustained periods of testing at least 4 times/day at appropriate intervals.
  Arms: Reinforcement for performing BG testing
Other: Standard of care — Subjects receive standard of care

SUMMARY:
The purpose of this project is to evaluate the efficacy of a behavioral economic intervention to improve self monitoring of blood glucose (SMBG) in adolescents and young adults with T1D. The intervention will reinforce patients for conducting SMBG, with escalating reinforcers provided when patients achieved sustained periods of testing at least 4 times/day at appropriate intervals. A 6-month trial will be conducted in which 60 patients will be randomized to: (1) standard care or (2) standard care plus the reinforcement intervention.

ELIGIBILITY:
Inclusion Criteria:

1. age 12-21 years old;
2. diagnosis of type 1 diabetes (T1D) >12 months via ADA guidelines
3. receiving diabetes treatment at Yale Pediatric Diabetes Clinic and not meeting clinical care guidelines
4. SMBG user with clinical recommendations to test >4 times/day and using a device that allows for remote uploading (e.g., Aviva, Contour, Freestyle, Lifescan, etc.; equipment for uploading will be provided);
5. access to a computer with internet for uploading and sending SMBG data;
6. access to a cell phone with text messaging capabilities and willing to text after SMBG testing and receive messages about reinforcement;
7. English speaking, able to read at >5th grade level, and pass an informed consent quiz; and adequate knowledge of insulin dosing and dietary recommendations for managing T1D.

Exclusion Criteria:

1. have a major psychiatric or neurocognitive disorder (e.g., severe learning impairment) that would inhibit participation;
2. have a major visual impairment;
3. have a significant other medical condition that impacts diabetes management (e.g., asthma, rheumatoid arthritis, or other condition that requires steroid treatment);
4. plan to switch insulin delivery mode (injection to pump or vice versa) in the next 12 months, or have recently switched;
5. are participating in another clinical trial.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2014-07; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
To determine if the reinforcement intervention increases SMBG testing. | 6 Months
  The number of SMBG tests will be assessed via glucometer uploads, and the proportion of days on which at least 4 tests occurred as well as the longest number of consecutive days on which SMBG tests occurred at frequencies of >4 times/day will be calculated. The hypothesis is that patients assigned to the reinforcement intervention will conduct more SMBG tests, have greater proportions of days with >4 tests, and have longer durations of appropriate testing frequencies than patients assigned to usual care.
To assess if the intervention reduces A1c | 6 months
  Patients randomized to the reinforcement intervention are expected to have greater decreases in A1c over time than patients assigned to usual care.

CONTACTS AND LOCATIONS:
Overall Officials: William Tamborlane, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No